CLINICAL TRIAL: NCT05455697
Title: Immunostart: Prephase Tafasitamab, Retifanlimab, and Rituximab (TRR), Followed by TRR With Standard Therapy for Previously Untreated Diffuse Large B-Cell Lymphoma
Brief Title: Tafasitamab, Retifanlimab, and Rituximab in Combination With Standard Therapy for the Treatment of Diffuse Large B-cell Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1122398; NCI-2022-04527 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RG1122398 (Other: Fred Hutch/University of Washington Cancer Consortium); 10946 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2022-06-17; First posted 2022-07-13 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Diffuse Large B-Cell Lymphoma; Grade 3b Follicular Lymphoma; High Grade B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Cyclophosphamide; Doxorubicin; Prednisone; Rituximab; Hyaluronoglucosaminidase; tafasitamab; Immunoglobulins; Disulfides; Vincristine; Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; X-Rays; polatuzumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (TRR, CHOP) (Experimental): PREPHASE THERAPY: Patients receive tafasitamab IV over 30 minutes on days 1, 8, and 15 of each cycle, rituximab and hyaluronidase human SC on day 1 of each cycle, and retifanlimab IV over 30 minutes on day 8 of each cycle. Treatment repeats every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity.
  COMBINATION THERAPY: After completion of prephase therapy or if patients progress during prephase therapy, patients receive tafasitamab IV over 30 minutes, retifanlimab IV over 30 minutes, rituximab and hyaluronidase human SC, cyclophosphamide IV, doxorubicin IV, and vincristine IV on day 1 of each cycle. Patients with an IPI score of 2-5 may receive polatuzumab vedotin IV in place of vincristine at investigator discretion. Patients also receive prednisone PO on days 1-5 of each cycle. Treatment repeats every 21 days for 4-6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Bone Marrow Biopsy; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone; Biological: Retifanlimab; Biological: Rituximab and Hyaluronidase Human; Biological: Tafasitamab; Drug: Vincristine; Procedure: Bone Marrow Aspiration; Procedure: Multigated Acquisition Scan; Other: Fludeoxyglucose F-18; Procedure: Positron Emission Tomography; Procedure: Computed Tomography; Procedure: Biospecimen Collection; Drug: Polatuzumab Vedotin

INTERVENTIONS:
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
Drug: Cyclophosphamide — Given IV
  Other Names: Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphanum; Cyclostine; Cytophosphane; Cytoxan; Fosfaseron; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Doxorubicin — Given IV
  Other Names: 14-Hydroxydaunomycin; 23214-92-8; Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Drug: Prednisone — Given PO
  Other Names: Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltra; Econosone; Lisacort; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Predicor; Predicorten; Prednicort; Prednilonga; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Biological: Retifanlimab — Given IV
  Other Names: 2226345-85-1; INCMGA 0012; INCMGA-0012; INCMGA00012; INCMGA0012; MGA 012; MGA-012; MGA012; Retifanlimab-dlwr; Zynyz
Biological: Rituximab and Hyaluronidase Human — Given SC
  Other Names: Rituxan Hycela; Rituximab Plus Hyaluronidase; Rituximab/Hyaluronidase; Rituximab/Hyaluronidase Human
Biological: Tafasitamab — Given IV
  Other Names: 1422527-84-1; Immunoglobulin; Anti-(Human Cd19 Antigen) (Human-mus musculus Monoclonal MOR00208 Heavy Chain); Disulfide with Human-mus musculus Monoclonal MOR00208 .Kappa.-chain,; Dimer; Monjuvi; MOR-00208; MOR00208; MOR208; Tafasitamab-cxix; XmAb5574
Drug: Vincristine — Given vincristine
  Other Names: 22-Oxovincaleukoblastine, 57-22-7; LEUROCRISTINE; VCR; Vincrystine
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide ventriculography; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Other: Fludeoxyglucose F-18 — Undergo FDG-PET/CT
  Other Names: 105851-17-0; 18FDG
Procedure: Positron Emission Tomography — Undergo FDG-PET
  Other Names: Medical Imaging; PET Scan; Positron Emission Tomography Scan
Procedure: Computed Tomography — Undergo FDG-CT
  Other Names: CAT Scan; Computed Axial Tomography; CT SCAN
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection
Drug: Polatuzumab Vedotin — Given IV
  Other Names: Antibody-Drug Conjugate DCDS4501A; Polivy

SUMMARY:
This phase I/II trial tests the safety of tafasitamab, retifanlimab, and rituximab (TRR) as a prephase treatment and in combination with standard therapy consisting off cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) or polatuzumab vedotin, cyclophosphamide, doxorubicin, and prednisone (PolaCHP) in patients with untreated diffuse large B-cell lymphoma. Tafasitamab, retifanlimab, and rituximab are monoclonal antibodies. Tafasitamab binds to a protein called CD19, which is found on B-cells (a type of white blood cell) and some types of cancer cells. Rituximab binds to a protein called CD20, which is also found on B-cells and some cancer cells. These monoclonal antibodies may help the immune system kill cancer cells. Immunotherapy with other monoclonal antibodies, such as retifanlimab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs, such as CHOP and PolaCHP, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving TRR in combination with CHOP or PolaCHP may kill more cancer cells.

DETAILED DESCRIPTION:
OUTLINE:

PREPHASE THERAPY: Patients receive tafasitamab intravenously (IV) over 30 minutes on days 1, 8, and 15 of each cycle, rituximab and hyaluronidase human subcutaneously (SC) on day 1 of each cycle, and retifanlimab IV over 30 minutes on day 8 of each cycle. Treatment repeats every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity.

COMBINATION THERAPY: After completion of prephase therapy or if patients progress during prephase therapy, patients receive tafasitamab IV over 30 minutes, retifanlimab IV over 30 minutes, rituximab and hyaluronidase human SC, cyclophosphamide IV, doxorubicin IV, and vincristine IV on day 1 of each cycle. Patients with an international prognostic index (IPI) score of 2-5 may receive polatuzumab vedotin IV in place of vincristine at investigator discretion. Patients also receive prednisone orally (PO) on days 1-5 of each cycle. Treatment repeats every 21 days for 4-6 cycles in the absence of disease progression or unacceptable toxicity.

Patients also undergo optional bone marrow biopsy and aspiration and multi-gated acquisition (MUGA) scan at screening, and fludeoxyglucose (FDG) positron emission tomography/computed tomography (PET/CT) scan and collection of blood and tissue samples throughout the trial.

After completion of study treatment, patients are followed up at 4-6 weeks, 12 weeks and then per routine care for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previously untreated diffuse large B cell lymphoma or grade 3B follicular lymphoma (of any stage). Patients may have de novo DLBCL, and /or any of the following:

  * Composite lymphomas, which include both diffuse DLBCL and another histology (most commonly follicular lymphoma) in the same lymph node,
  * Transformed lymphoma with DLBCL histology, as long as the patient has not received prior therapy for lymphoma,
  * Discordant presentations, such as DLBCL in a lymph node and low-grade lymphoma such as follicular lymphoma in the bone marrow, and
  * High grade B-cell lymphoma (including "double hit" lymphomas or high grade B-cell lymphoma-not otherwise specified [HGBCL-NOS]) is permitted if the patient is not eligible for or declines intensive therapy
* Be willing and able to provide written informed consent/assent for the trial
* Be >= 18 years of age on day of signing informed consent
* Have measurable disease, including at least 1 nodal site measuring 1.5 cm or 1 extranodal site measuring 1.0 cm in longest dimension on computed tomography (CT) or fludeoxyglucose F-18-positron emission tomography (FDG-PET)
* Have a performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) performance scale (PS)
* Absolute neutrophil count (ANC) >= 1,000/mcL except in case of marrow infiltration by lymphoma
* Platelets >= 75,000/mcL except in cases of marrow infiltration by lymphoma
* Serum creatinine clearance (CrCl) must be >= 30 mL/minute either measured or calculated using a standard Cockcroft and Gault formula

  * Creatinine clearance should be calculated per institutional standard
* Serum total bilirubin =< 1.5 x upper limit of normal (ULN) unless secondary to Gilbert's syndrome or documented liver involvement by lymphoma. Patients with Gilbert's syndrome or documented liver involvement by lymphoma may be included if their total bilirubin is =< 5 x ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN OR =< 5 x ULN for subjects with liver metastases
* Left ventricular ejection fraction of >= 45%, assessed by echocardiography or cardiac multi-gated acquisition (MUGA) scan
* Female subjects of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control, be surgically sterile, or abstain from heterosexual activity starting with the first dose of study therapy and for 180 days after the last dose of study medication. Female subjects of childbearing potential must also agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the trial and for 180 days after receiving the last dose of study therapy. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use 2 methods of contraception starting with the first dose of study therapy and for 180 days after the last dose of study therapy

Exclusion Criteria:

* Is currently participating in a study and receiving an investigational agent or is using an investigational device within 4 weeks of the first dose of treatment
* Requires systemic corticosteroids in excess of > 10 mg/day of prednisone or equivalent. Exceptions:

  * Physiologic corticosteroid replacement therapy at doses =< 10 mg/day of prednisone or equivalent for adrenal or pituitary insufficiency and in the absence of active autoimmune disease is permitted
  * Participants with asthma that require intermittent use of bronchodilators, inhaled steroids, or local steroid injections may participate
  * Participants using topical, ocular, intra-articular, or intranasal steroids (with minimal systemic absorption) may participate
  * Brief courses of corticosteroids for prophylaxis (e.g., contrast dye allergy) or prephase steroids for disease control, given for up to 7 days, are permitted
  * Steroids required for management of immune-related adverse events after initiation of study therapy are permitted
* Has a diagnosis of immunodeficiency
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include resected cutaneous neoplasms, in situ cancer, or any neoplasm not requiring therapy or with a life expectancy exceeding 3 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Evidence of interstitial lung disease, history of interstitial lung disease, or active, noninfectious pneumonitis
* Has an active infection requiring intravenous antibiotic therapy at the time of start of study therapy
* History of organ transplant, including allogeneic stem cell transplantation
* Has received a live vaccine within 28 days of the planned start of study drug

  * Note: Examples of live vaccines include but are not limited to intranasal influenza, measles, mumps, rubella, chicken pox/zoster, yellow fever, rabies, BCG, and typhoid vaccine
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 180 days after the last dose of trial treatment
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies), unless controlled on therapy and CD4 count is > 200/uL
* Has known active Hepatitis B (e.g., hepatitis B virus surface antigen [HBsAg] reactive or hepatitis B virus [HBV] deoxyribonucleic acid [DNA] detectable) or Hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2027-01-05 (Estimated); Study Completion 2027-07-06 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity rate | From treatment start to end of cycle 3 (each cycle is 3 weeks)
  Statistical analysis will entail descriptive statistics of adverse event rates. Will build a Cox proportional hazard model for univariate analysis and multivariable analysis if applicable. Correlative studies may incorporate t-test and linear regression for continuous variables, Chi-squared test and logistic regression for categorical variables will be used, if applicable.

SECONDARY OUTCOMES:
Overall response rate | Up to 5 years
  Will build a Cox proportional hazard model for univariate analysis and multivariable analysis if applicable. Correlative studies may incorporate t-test and linear regression for continuous variables, Chi-squared test and logistic regression for categorical variables will be used, if applicable.
Progression-free survival | Time from start of trial therapy until relapse or progression, non-protocol re-treatment of lymphoma, or death as a result of any cause, assessed up to 5 years
  Time-to-event analyses for progression-free survival will be conducted using the Kaplan-Meier method and log-rank test. Will build a Cox proportional hazard model for univariate analysis and multivariable analysis if applicable. Correlative studies may incorporate t-test and linear regression for continuous variables, Chi-squared test and logistic regression for categorical variables will be used, if applicable.
Overall survival | From start of trial therapy to death from any cause, assessed up to 5 years
  Time-to-event analyses for overall survival will be conducted using the Kaplan-Meier method and log-rank test. Will build a Cox proportional hazard model for univariate analysis and multivariable analysis if applicable. Correlative studies may incorporate t-test and linear regression for continuous variables, Chi-squared test and logistic regression for categorical variables will be used, if applicable.
Proportion completing prephase | Up to 5 years
  Will build a Cox proportional hazard model for univariate analysis and multivariable analysis if applicable. Correlative studies may incorporate t-test and linear regression for continuous variables, Chi-squared test and logistic regression for categorical variables will be used, if applicable.
Relative dose intensity of doxorubicin and cylcophosphamide during combination therapy | Up to 5 years
  Relative dose intensity for doxorubicin and cyclophosphamide will be calculated as follows:
  * Standard dose intensity (SDI): (Standard total dose, in mg/m2 )/(standard time to complete chemotherapy, in days
  * Delivered dose intensity (DDI): (Delivered total dose, in mg/m2)/(actual time to complete chemotherapy, in days)
  * Relative dose intensity: DDI/SDI x 100% Will build a Cox proportional hazard model for univariate analysis and multivariable analysis if applicable. Correlative studies may incorporate t-test and linear regression for continuous variables, Chi-squared test and logistic regression for categorical variables will be used, if applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D. Smith, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No